CLINICAL TRIAL: NCT01586247
Title: A Double-blind, Placebo-controlled, Randomized Crossover Study of a Prebiotic (Galacto-oligosaccharides, GOS), Probiotic (B.Lactis, BI07) and Synbiotic (GOS + BI07) on the Gut Microbiota and Immune Response of Older Volunteers
Brief Title: The Effect of a Prebiotic, Probiotic and Synbiotic on the Gut Microbiota and Immune Response of Older Volunteers (GOS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: Danisco (Industry)
Responsible Party: Principal Investigator, Caroline Childs, Post doctoral research fellow, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 07/47
Record Dates: First submitted 2012-04-19; First posted 2012-04-26 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Gut Microbiota; Immune Function
MeSH Terms: interventions — Synbiotics; Prebiotics; Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Synbiotic (Experimental): 8g/day gluco-oligosaccharide + 109 CFU/day B. lactis BI07
  Interventions: Dietary Supplement: Synbiotic
- Placebo (Experimental): 8g/day maltodextrin
  Interventions: Dietary Supplement: Placebo
- Prebiotic (Experimental): 8g/day galacto-oligosaccharides (GOS)
  Interventions: Dietary Supplement: Prebiotic
- Probiotic (Experimental): 109 CFU/day B. lactis BI07
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Synbiotic — 8g/day galacto-oligosaccharide + 10^9 CFU/day B.lactis
  Other Names: GOS Bi-07
  Arms: Synbiotic
Dietary Supplement: Placebo — 8g/day maltodextrin
  Arms: Placebo
Dietary Supplement: Prebiotic — 8g/day galacto-oligosaccharide
  Other Names: GOS
  Arms: Prebiotic
Dietary Supplement: Probiotic — 10^9 CFU/day B.lactis
  Other Names: Bi-07
  Arms: Probiotic

SUMMARY:
Healthy older volunteers will be recruited to a study where they will be given four different treatments over a 28 week period. These treatments include: a prebiotic, a probiotic, a synbiotic (prebiotic + probiotic) and a placebo. Faecal samples, blood and saliva will be collected and analysed for changes in faecal microbial populations and selected immune responses.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the effect of GOS (administered at 8g/day), B. lactis BI07 (administered at 109 CFU/day) and the synbiotic (8g/day of GOS and 109 CFU/day of B. lactis BI07) on the human gut microbiota.

A double-blind, placebo-controlled, randomized crossover study will be conducted in 40 healthy older (≥60 years of age) volunteers. The placebo will consist of maltodextrin (a food grade ingredient, administered at 8g/day).

Changes in the gut microbiota will be determined by measuring bacterial population levels in human faeces using 16S rRNA targeted oligonucleotide probes and fluorescence in situ hybridisation. Faecal pH will be measured and the production of short chain fatty acids (SCFA) will be analysed and quantified using high performance liquid chromatography (HPLC).

The secondary objective of this study is to examine the effect on cellular immune function. This will be achieved by investigating phagocytosis activity, natural killer cells which are CD4+, CD8+, CD25+ and CD2+ and CD3+ subsets, the marker of T-cell maturation period., salivary IgA levels, inflammatory markers (plasma - tumour necrosis factor (TNF), IL6, IL1, chemokines and soluble adhesion molecules).

ELIGIBILITY:
Inclusion Criteria:

* a signed consent form,
* age >60 years
* good general health
* not in the residential care.

Exclusion Criteria:

* evidence of physical or mental disease
* planned major surgery
* use of antibiotics within the previous six months

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-03; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Changes to the gut microbiota | Baseline and after 21d treatment
  The primary objective of this study is to determine the effect of GOS (administered at 8g/day), B. lactis BI07 (administered at 109 CFU/day) and the synbiotic (8g/day of GOS and 109 CFU/day of B. lactis BI07) on the human gut microbiota. Changes in the gut microbiota will be determined by measuring bacterial population levels in human faeces using 16S rRNA targeted oligonucleotide probes and fluorescence in situ hybridisation. Faecal pH will be measured and the production of short chain fatty acids (SCFA) will be analysed and quantified using high performance liquid chromatography (HPLC).

SECONDARY OUTCOMES:
Immune function | Baseline and after 21d treatment
  To examine the effect of GOS (administered at 8g/day), B. lactis BI07 (administered at 109 CFU/day) and the synbiotic (8g/day of GOS and 109 CFU/day of B. lactis BI07 ) on cellular immune function in 40 healthy older (≥60 years of age) volunteers. This will be achieved by investigating phagocytosis activity, natural killer cells which are CD4+, CD8+, CD25+ and CD2+ and CD3+ subsets, the marker of T-cell maturation period., salivary IgA levels, inflammatory markers (plasma - tumour necrosis factor (TNF), IL6, IL1, chemokines and soluble adhesion molecules).

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Rastall, Principal Investigator — University of Reading
Locations (1):
- University of Reading, Reading, Berkshire, United Kingdom